CLINICAL TRIAL: NCT01440764
Title: Aerosol Inhalation Treatment for Dyspnea
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Robert Banzett, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2011-P-000027/1; R01NR012009 (NIH)
Record Dates: First submitted 2011-09-23; First posted 2011-09-27 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Healthy; Dyspnea
Keywords: dyspnea; Laboratory model of dyspnea in healthy subjects
MeSH Terms: conditions — Dyspnea | interventions — Furosemide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- F(40), then Saline, then IV.F (Experimental): On Test Day 1, participants received Aerosol Furosemide 40mg in 4ml saline by inhalation for 5-10 minutes.
  On Test Day 2 (at least 24 hours after Test Day 1), participants received Aerosol Saline 4ml by inhalation for 5-10 minutes.
  On Test Day 3 (at least 24 hours after Test Day 2), participants received Furosemide 15 mg diluted in 10 ml of saline by intravenous delivery for 5 minutes.
  Interventions: Drug: Furosemide; Drug: Saline
- IV.F, then F(40), then Saline (Experimental): On Test Day 1, participants received Furosemide 15 mg diluted in 10 ml of saline by intravenous delivery for 5 minutes.
  On Test Day 2 (at least 24 hours after Test Day 1), participants received Aerosol Furosemide 40mg in 4ml saline by inhalation for 5-10 minutes.
  On Test Day 3 (at least 24 hours after Test Day 2), participants received Aerosol Saline 4ml by inhalation for 5-10 minutes.
  Interventions: Drug: Furosemide; Drug: Saline
- Saline, then F(40), then IV.F (Experimental): On Test Day 1, participants received Aerosol Saline 4ml by inhalation for 5-10 minutes.
  On Test Day 2 (at least 24 hours after Test Day 3), participants received Aerosol Furosemide 40mg in 4ml saline by inhalation for 5-10 minutes.
  On Test Day 3 (at least 24 hours after Test Day 2), participants received Furosemide 15 mg diluted in 10 ml of saline by intravenous delivery for 5 minutes.
  Interventions: Drug: Furosemide; Drug: Saline
- F(80), then Saline, then Saline (Experimental): On Test Day 1, participants received Aerosol Furosemide 80mg in 8ml saline by inhalation for 5-10 minutes.
  On Test Day 2 (at least 24 hours after Test Day 1), participants received Aerosol Saline 8ml by inhalation for 5-10 minutes.
  On Test Day 3 (at least 24 hours after Test Day 2), participants received Aerosol Saline 8ml by inhalation for 5-10 minutes.
  Interventions: Drug: Furosemide; Drug: Saline
- Saline, then F(80), then Saline (Experimental): On Test Day 1, participants received Aerosol Saline 8ml by inhalation for 5-10 minutes.
  On Test Day 2 (at least 24 hours after Test Day 1), participants received Aerosol Furosemide 80mg in 8ml saline by inhalation for 5-10 minutes.
  On Test Day 3 (at least 24 hours after Test Day 2), participants received Aerosol Saline 8ml by inhalation for 5-10 minutes.
  Interventions: Drug: Furosemide; Drug: Saline
- Saline, then Saline, then F(80) (Experimental): On Test Day 1, participants received Aerosol Saline 8ml by inhalation for 5-10 minutes.
  On Test Day 2 (at least 24 hours after Test Day 1), participants received Aerosol Saline 8ml by inhalation for 5-10 minutes.
  On Test Day 3 (at least 24 hours after Test Day 2), participants received Aerosol Furosemide 80mg in 8ml saline by inhalation for 5-10 minutes.
  Interventions: Drug: Furosemide; Drug: Saline

INTERVENTIONS:
Drug: Furosemide
  Other Names: Lasix
Drug: Saline

SUMMARY:
The purpose of this protocol is to develop and test optimal delivery of aerosol furosemide, a treatment that has the potential to significantly improve symptom management and enhance the quality of care for patients with intractable dyspnea.

DETAILED DESCRIPTION:
This is study of aerosol treatment in a laboratory model of dyspnea in healthy subjects. This study is the first in a series of studies that will include investigation of a second dose in the laboratory and investigation of the treatment effect in hospitalized patients with refractory dyspnea. The outcome of this first study will determine the details of protocol for the succeeding studies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Unstable heart or circulation disease
* Stroke
* Seizure disorder
* Severe migraine headaches
* Liver or kidney disease
* Adrenal gland problem (Pheochromocytoma)
* Nerve problems that may affect your breathing sensation
* Brain cancer
* Drug or alcohol problem
* Systemic lupus erythematosis (SLE)
* High levels of depression, panic disorder, or other significant mental health problems
* Serious ongoing pain
* Pregnant
* Under 18 years old
* Not Fluent in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2016-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B Banzett, PhD, Principal Investigator — Beth Israel Deaconess Hospital
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Banzett RB, Adams L, O'Donnell CR, Gilman SA, Lansing RW, Schwartzstein RM. Using laboratory models to test treatment: morphine reduces dyspnea and hypercapnic ventilatory response. Am J Respir Crit Care Med. 2011 Oct 15;184(8):920-7. doi: 10.1164/rccm.201101-0005OC. Epub 2011 Jul 21. PMID 21778294

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a crossover study of a total of 24 people.
Groups:
- Saline, Then F(40), Then IV.F: On Test Day 1, participants received Aerosol Saline 4ml by inhalation for 5-10 minutes.
  On Test Day 2 (at least 24 hours after Test Day 1), participants received Aerosol Furosemide 40mg in 4ml saline by inhalation for 5-10 minutes.
  On Test Day 3 (at least 24 hours after Test Day 2), participants received Furosemide 15 mg diluted in 10 ml of saline by intravenous delivery for 5 minutes.
- Saline, Then F(80), Then IV.F: On Test Day 1, participants received Aerosol Furosemide 80mg in 8ml saline by inhalation for 5-10 minutes.
  On Test Day 2 (at least 24 hours after Test Day 1), participants received Aerosol Saline 8ml by inhalation for 5-10 minutes.
  On Test Day 3 (at least 24 hours after Test Day 2), participants received Furosemide 15 mg diluted in 10 ml of saline by intravenous delivery for 5 minutes.
Period: Test Day 1
Arm/Group | F(40), Then Saline, Then IV.F | IV.F, Then F(40), Then Saline | Saline, Then F(40), Then IV.F | Saline, Then F(80), Then IV.F | F(80), Then Saline, Then Saline | Saline, Then F(80), Then Saline | Saline, Then Saline, Then F(80)
Started | 4 | 2 | 6 | 1 | 3 | 5 | 3
Completed | 4 | 2 | 6 | 1 | 3 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Test Day 2
Arm/Group | F(40), Then Saline, Then IV.F | IV.F, Then F(40), Then Saline | Saline, Then F(40), Then IV.F | Saline, Then F(80), Then IV.F | F(80), Then Saline, Then Saline | Saline, Then F(80), Then Saline | Saline, Then Saline, Then F(80)
Started | 3 (Following Test Day 1, 1 subject withdrew from the study before beginning Test Day 2.) | 2 | 6 | 1 | 3 | 5 | 3
Completed | 3 | 2 | 6 | 1 | 3 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Test Day 3
Arm/Group | F(40), Then Saline, Then IV.F | IV.F, Then F(40), Then Saline | Saline, Then F(40), Then IV.F | Saline, Then F(80), Then IV.F | F(80), Then Saline, Then Saline | Saline, Then F(80), Then Saline | Saline, Then Saline, Then F(80)
Started | 3 | 2 | 6 | 1 | 3 | 5 | 3
Completed | 3 | 2 | 6 | 1 | 3 | 5 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- F(40) Participants: Participants who consented to participate in the study and receive the Aerosol Furosemide (40mg/4ml solution of Saline), Aerosol Saline (4ml), and IV Furosemide (15mg/8ml Saline) Interventions in any sequence.
- F(80) Participants: Participants who consented to participate in the study and receive the Aerosol Furosemide (80mg/8ml solution of Saline) and two Aerosol Saline (8ml) Interventions in any sequence or receive the Aerosol Furosemide (80mg/8ml solution of Saline), Aerosol Saline (8ml), and IV Furosemide (15mg/8ml Saline) Interventions in any sequence.
- Total: Total of all reporting groups
Arm/Group | F(40) Participants | F(80) Participants | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.25 (12.65) | 23.58 (4.42) | 27.42 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 10 | 13
  Male | 9 | 2 | 11
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Subject Rating of Breathing Discomfort (Dyspnea)
Description: Change in breathing discomfort (dyspnea) rating at benchmark PETCO2 using a visual analog scale. The change in breathing discomfort is expressed as units on a 0% to 100% continuous scale, where higher values represent more dyspnea. The change is represented as the rating of breathing discomfort after the intervention minus the rating of breathing discomfort before the intervention.
Time Frame: The breathing discomfort ratings were taken as an average of all ratings during runs before intervention and the first two runs after intervention. The 1st and 2nd post-runs began (on average) 12 minutes and 49 minute after intervention, respectively.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Aerosol Furosemide (40 mg): Participants who received Aerosol Furosemide 40mg in 4ml saline by inhalation for 5-10 minutes on a single test day and met quality control.
  Of the 12 participants who consented to receive this intervention, all 12 participants received the intervention and completed the study day. However, it was later discovered that 1 subject had used cannabis recently and their information was discarded. Therefore, this analysis includes only the 11 subjects who met quality control.
- Aerosol Saline (4 ml): Participants who received Aerosol Saline (4ml) by inhalation for 5-10 minutes on a single test day and met quality control.
  Of the 12 participants who consented to receive this intervention, only 11 participants received the intervention and completed the study day (one withdrew before starting this intervention).
  Additionally, it was later discovered that 1 subject had used cannabis recently and their data was discarded.
  Therefore, this analysis includes only the 10 subjects who met quality control.
- IV Furosemide: Participants who received Furosemide 15 mg diluted in 10 ml of saline by intravenous delivery for 5 minutes on 1 test day and met quality control.
  Of the 13 participants who consented to receive this intervention, only 12 participants received the intervention and completed the study day (one withdrew before starting this intervention).
  Additionally, it was later discovered that 1 subject had used cannabis recently and their data was discarded. Also, 1 subject's data did not meet quality control and was excluded.
  Therefore, this analysis includes only the 10 subjects who met quality control.
- Aerosol Furosemide (80mg): Participants who received Aerosol Furosemide 80mg in 8ml saline by inhalation for 5-10 minutes on 1 test day and met quality control.
  12 participants who consented to receive this intervention received the intervention and completed the study day. However, 1 subject's physiological data did not meet quality control and was discarded. Therefore, this analysis includes only the 11 subjects who met quality control.
- Aerosol Saline (8 ml): Aerosol Saline 8ml by inhalation for 5-10 minutes on 2 test days and met quality control.
  12 participants who consented to receive this intervention received the intervention and completed the study day. However, 1 subject's physiological data did not meet quality control and was discarded. Therefore, this analysis includes only the 11 subjects who met quality control.
Arm/Group | Aerosol Furosemide (40 mg) | Aerosol Saline (4 ml) | IV Furosemide | Aerosol Furosemide (80mg) | Aerosol Saline (8 ml)
Number analyzed (Participants) | 11 | 10 | 10 | 11 | 11
units on a scale | 20 (13) | 20 (10) | 16 (13) | 17 (3) | 13 (4)
Statistical Analysis 1: Comparison: Aerosol Furosemide (40 mg) vs Aerosol Saline (4 ml); Test type: Superiority; p = 0.99, t-test, 2 sided — a priori threshold for significance was 0.05. Not corrected for multiple comparisons. This p-value describes the a priori analysis of comparing the furosemide test result to the saline test result
Statistical Analysis 2: Comparison: Aerosol Furosemide (80mg) vs Aerosol Saline (8 ml); Test type: Superiority; p = 0.32, t-test, 2 sided — a priori threshold for significance was 0.05. Not corrected for multiple comparisons. Thes p-value describes the a priori analysis of comparing the response to furosemide to the mean response to saline

2. Secondary Outcome: Multidimensional Dyspnea Profile
Description: Characterization of subject's response to laboratory dyspnea model. Data are from a baseline pre-treatment test on the first drug or placebo treatment day for the subjects used in the main analysis. Subjects were asked to complete the MDP with reference to the last 30 sec of each run. To weigh subjects equally, we selected one run from each subject: the first run that terminated in a rating of overall breathing discomfort (A1) of 50 to 90% of full scale. The units of measurement are expressed as units on a 0 to 10 scale measuring intensity of a given quality, with higher values indicating greater intensity and 10 representing maximum perceived intensity.
Time Frame: Measured before intervention
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Aerosol Furosemide (80mg): Participants who received Aerosol Furosemide 80mg in 8ml saline by inhalation for 5-10 minutes on a single test day and met quality control.
  Of the 12 participants who consented to receive this intervention, all 12 participants received the intervention and completed the study day. However, it was later discovered that 1 subject's data did not pass a priori requirements for quality control and the subject's data was excluded. Therefore, this analysis includes only the 11 subjects who met quality control.
Arm/Group | Aerosol Furosemide (40 mg) | Aerosol Furosemide (80mg)
Number analyzed (Participants) | 11 | 11
units on a scale
  A1 (overall breathing discomfort) | 8.0 (0.2) | 6.4 (0.4)
  Muscle Work | 5.5 (0.8) | 2.5 (0.7)
  Air hunger | 7.4 (0.5) | 6.2 (0.8)
  Tightness | 3.3 (0.8) | 2.6 (0.9)
  Mental effort | 6.3 (0.7) | 3.6 (0.9)
  Breathing a lot | 4.0 (0.9) | 1.5 (0.7)
  Depressed | 0.3 (0.2) | 0.0 (0.0)
  Anxious | 3.7 (0.7) | 2.9 (0.6)
  Frustrated | 1.6 (0.7) | 1.6 (0.6)
  Angry | 0.9 (0.5) | 0.2 (0.2)
  Afraid | 1.1 (0.4) | 1.2 (0.4)

3. Secondary Outcome: Urine Output
Description: Diuresis is an expected effect of furosemide. To the extent that aerosol furosemide is absorbed into the blood, diuresis is an expected 'side effect' of this treatment
Time Frame: Cumulative urine output 1 hour after intervention
Measure: Mean (Standard Deviation); unit: ml of urine
Groups:
- Aerosol Furosemide (40 mg): Aerosol Furosemide 40mg in 4ml saline by inhalation for 5-10 minutes on 1 test day.
  To be compared to Aerosol Saline (4ml) Arm and IV Furosemide Arm.
  Furosemide
- Aerosol Furosemide (80mg): Aerosol Furosemide 80mg in 8ml saline by inhalation for 5-10 minutes on 1 test day.
  To be compared to Aerosol Saline (8ml) Arm.
  Furosemide
- Aerosol Saline (4 ml): Aerosol Saline 4ml by inhalation for 5-10 minutes on 1 test day.
  To be compared to Aerosol Furosemide (40mg) Arm and IV Furosemide Arm.
  Saline
- Aerosol Saline (8 ml): Aerosol Saline 8ml by inhalation for 5-10 minutes on 2 test days.
  To be compared to Aerosol Furosemide (80mg) Arm.
  Saline
- IV Furosemide: Furosemide 15 mg diluted in 10 ml of saline by intravenous delivery for 5 minutes on 1 test day.
  To be compared to Aerosol Furosemide (40mg) Arm and Aerosol Saline (4 ml) Arm.
  Furosemide
Arm/Group | Aerosol Furosemide (40 mg) | Aerosol Furosemide (80mg) | Aerosol Saline (4 ml) | Aerosol Saline (8 ml) | IV Furosemide
Number analyzed (Participants) | 12 | 11 | 10 | 11 | 11
ml of urine | 1069 (435) | 1320 (394) | 500 (264) | 474 (146) | 1556 (435)
Statistical Analysis 1: Comparison: Aerosol Furosemide (40 mg) vs Aerosol Saline (4 ml); Test type: Superiority; p = .0006, t-test, 2 sided — a priori threshold for statistical significance was 0.05. Not adjusted for multiple comparisons
Statistical Analysis 2: Comparison: Aerosol Furosemide (80mg) vs Aerosol Saline (8 ml); Test type: Superiority; p = .00001, t-test, 2 sided — a priori threshold for statistical significance was 0.05. Not adjusted for multiple comparisons
Statistical Analysis 3: Comparison: Aerosol Saline (4 ml) vs IV Furosemide; Test type: Superiority; p = .0000002, t-test, 2 sided — a priori threshold for significance was 0.05. Not adjusted for multiple comparisons

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Aerosol Furosemide (40 mg): Any subject who received Aerosol Furosemide 40mg in 4ml saline by inhalation for 5-10 minutes on 1 test day.
- Aerosol Furosemide (80mg): Any subject who received Aerosol Furosemide 80mg in 8ml saline by inhalation for 5-10 minutes on 1 test day.
- Aerosol Saline (4 ml): Any subject who received Aerosol Saline 4ml by inhalation for 5-10 minutes on 1 test day.
- Aerosol Saline (8 ml): Any subject who received Aerosol Saline 8ml by inhalation for 5-10 minutes on 2 test days.
- IV Furosemide: Any subject who received Furosemide 15 mg diluted in 10 ml of saline by intravenous delivery for 5 minutes on 1 test day.
Arm/Group | Aerosol Furosemide (40 mg) | Aerosol Furosemide (80mg) | Aerosol Saline (4 ml) | Aerosol Saline (8 ml) | IV Furosemide
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/11 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/11 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/11 | 0/11 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No